CLINICAL TRIAL: NCT01966159
Title: EVOLVE China: A Prospective, Multicenter Trial to Assess the Safety and Effectiveness of the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System) for the Treatment of Atherosclerotic Lesion(s)
Brief Title: The EVOLVE China Clinical Trial
Acronym: EVOLVE-CHINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2279
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYNERGY Investigational Device (Experimental): SYNERGY Stent System
  Interventions: Device: SYNERGY Investigational Device
- PE Plus Investigational Device (Active Comparator): PE Plus Stent System
  Interventions: Device: PE Plus Investigational Device

INTERVENTIONS:
Device: SYNERGY Investigational Device — percutaneous coronary intervention
  Arms: SYNERGY Investigational Device
Device: PE Plus Investigational Device — percutaneous coronary intervention
  Arms: PE Plus Investigational Device

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the SYNERGY™ Coronary Stent System for the treatment of subjects with atherosclerotic lesion(s) ≤ 34 mm in length (by visual estimate) in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate)

DETAILED DESCRIPTION:
The EVOLVE China clinical trial is designed to assess the safety and effectiveness of the SYNERGY™ Everolimus-Eluting Platinum Chromium Coronary Stent System for the treatment of subjects with atherosclerotic lesion(s) in native coronary arteries in China. The SYNERGY™ Stent System (Boston Scientific Corporation [BSC Corporation], Natick, Massachusetts, United States) is based on the well characterized Element™ stent platform and utilizes a bioabsorbable poly(DL-lactide-co-glycolide) (PLGA) polymer to deliver everolimus.

While SYNERGY is a new generation DES, the safety and effectiveness of the Element stent platform in combination with everolimus in the form of the PROMUS Element stent has been established in the PLATINUM Clinical Trial Program.The PROMUS Element Plus stent (control device) uses the same stent platform as PROMUS Element stent with a modified balloon component on the Stent Delivery System to improve overall system deliverability. In addition, the previous version of the SYNERGY stent, the SYNERGY First Human Use stent (SYNERGY FHU stent) has been investigated in the EVOLVE FHU trial which has completed its primary endpoint and demonstrated comparable safety and efficacy profile of SYNERGY FHU to PROMUS Element up to 1-year follow-up (28). SYNERGY has been approved by CE Mark.

ELIGIBILITY:
Inclusion Criteria:

* CI1. Subject must be 18 -75 years of age
* CI2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* CI3. Subject is eligible for percutaneous coronary intervention (PCI)
* CI4. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
* CI5. Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
* CI6. Subject is willing to comply with all protocol-required follow-up evaluation
* CI7. Subject has a left ventricular ejection fraction (LVEF) >30% as measured within 60 days prior to enrollment
* AI1. Target lesion(s) must be de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm
* AI2. Target lesion(s) length must be ≤34 mm (by visual estimate)
* AI3. Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following: stenosis ≥70%, abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure
* AI4. Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)
* AI5. The first lesion treated must be successfully predilated/pretreated

Exclusion Criteria:

* CE1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI .
* CE2. Subject with unstable angina or recent MI (within 1 week) must have CK/CK-MB or troponin documented prior to the procedure and are excluded if any of the following criteria are met at the time of the index procedure:

  * If CK MB >2× upper limit of normal (ULN), the subject is excluded regardless of the CK Total.
  * If CK Total >2× ULN, either CK-MB or troponin must be drawn and the subject is excluded if either CK-MB or troponin is abnormal.
  * If neither CK Total or CK MB is drawn but troponin is, the subject is excluded if troponin >1× ULN and the subject has at least one of the following:

    * Subject has ischemic symptoms and ECG changes indicative of ongoing ischemia (e.g., >1 mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB])
    * Development of pathological Q waves in the ECG or
    * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality
* CE3. Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, or intractable ventricular arrhythmias or ongoing intractable angina
* CE4. Subject has received an organ transplant or is on a waiting list for an organ transplant
* CE5. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* CE6. Planned PCI or CABG after the index procedure
* CE7. Subject has a known allergy to the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, clopidogrel, or aspirin) and contrast (that cannot be adequately premedicated)
* CE8. Subject has a known condition(s) of the following (as assessed from the time of screening through the day of index procedure):

  * Other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* CE9. Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, Coumadin) for indications other than acute coronary syndrome
* CE10. Subject with out of range complete blood count (CBC) values that are determined by the study physician to be clinically significant.
* CE11. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* CE12. Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* CE13. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* CE14. Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* CE15. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* CE16. Subject has signs or symptoms of active heart failure (i.e., NYHA class IV) at the time of the index procedure
* CE17. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* CE18. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* CE19. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* CE20. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* CE21. Target vessel has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure
* AE1. Planned treatment of more than 2 lesions
* AE2. Planned treatment of lesions in more than 2 major epicardial vessels
* AE3. Planned treatment of a single lesion with more than 1 stent Note: Planned use of 2 overlapping stents will be allowed in subjects randomized to PROMUS Element Plus where lesion length is ≥28 mm and 2.25 mm stents are used.
* AE4. Target lesion meets any of the following criteria:

  * Left main location
  * Located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate
  * Located within a saphenous vein graft or an arterial graft
  * Will be accessed via a saphenous vein graft or an arterial graft
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
  * Thrombus, or possible thrombus, present in the target vessel
  * Excessive tortuosity proximal to or within the lesion
  * Excessive angulation proximal to or within the lesion
  * Target lesion and/or the target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Involves a side branch ≥2.0 mm in diameter by visual estimate or a side branch <2.0 mm in diameter by visual estimate which requires treatment
* AE5. Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
* AE6. Target lesion(s) is restenostic from a previous stent implantation or study stent would overlap with a previous stent
* AE7. Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* AE8. Subject has protected left main coronary artery disease (>50% diameter stenosis in the LMCA with bypass graft(s) to the left coronary artery) and a target lesion in the LAD or LCX

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Dr., Principal Investigator — Shenyang Northern Hospital (The General Hospital of Shenyang Military Region)
Locations (14):
- China (14):
  - Beijing Affiliated Hospital of Armed Police Medical College, Beijing
  - Beijing Hospital of the Ministry of Health, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Daqing General Oil Field Hospital, Daqing
  - Guangdong Cardiovascular Institute of Guangdong Provincial Hospital, Guangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - Shengjing Hospital of China Medical University, Shengyang
  - Shenyang Northern Hospital (The General Hospital of Shenyang Military Region), Shenyang
  - TEDA International Cardiovascular Hospital, Tianjin
  - Logistics University of PAPF Affiliated Hospital, Tianjing
  - Wuhan Asia Heart Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Xijing Hospital, Fourth Military Medical University, Xi'an

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 412 subjects have enrolled and finished at 07Jul2014
Groups:
- SYNERGY Investigational Device (Test): SYNERGY Investigational Device (Test): percutaneous coronary intervention
- PROMUS Element Plus Investigational Device (Control): PROMUS Element Plus Investigational Device (Control): percutaneous coronary intervention
Period: Overall Study
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control)
Started | 205 | 207
Completed | 205 | 207
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control) | Total
Number analyzed (Participants) | 205 | 207 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.41 (8.76) | 57.89 (9.19) | 58.15 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 143 | 148 | 291
Region of Enrollment [Number; unit: participants]
  China | 205 | 207 | 412

OUTCOME MEASURES:

1. Primary Outcome: The In-stent Late Loss Measured by Quantitative Coronary Angiography
Time Frame: at 9 months post-index procedure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control)
Number analyzed (Participants) | 205 | 207
mm | 0.20 (0.33) | 0.17 (0.38)

2. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Description: Target lesion revascularization is any ischemia-driven repeat percutaneous intervention, to improve blood flow, of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 12 months post-index procedure
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control)
Number analyzed (Participants) | 205 | 207
percentage of participants | 2.0 | 2.9

3. Other Pre Specified Outcome: Target Lesion Failure (TLF) Rate
Description: Target lesion failure is any ischemia-driven revascularization of the target lesion, MI (Q-wave and non-Q-wave) related to the target vessel, or (cardiac) death.
Time Frame: 12 months post-index procedure
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control)
Number analyzed (Participants) | 205 | 207
percentage of participants | 4.0 | 4.4

ADVERSE EVENTS:
Time Frame: 12 month
Arm/Group | SYNERGY Investigational Device (Test) | PROMUS Element Plus Investigational Device (Control)
Serious Adverse Events (participants affected / at risk) | 38/205 | 27/207
Other Adverse Events (participants affected / at risk) | 66/205 | 60/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Investigational Device (Test) (N=205) | PROMUS Element Plus Investigational Device (Control) (N=207)
Angina unstable (Cardiac disorders) | 5 (7) | 5 (5)
chest discomfort (General disorders) | 2 (3) | 0 (0)
cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
aortic intramural haematoma (Vascular disorders) | 1 (1) | 1 (1)
coronary artery stenosis (Cardiac disorders) | 3 (3) | 3 (3)
mycardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
coronary artery dissection (Cardiac disorders) | 2 (2) | 2 (2)
coronary artery disease (Cardiac disorders) | 1 (1) | 4 (4)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
atriventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
ventricular arthythmia (Cardiac disorders) | 1 (1) | 0 (0)
coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
oedema peripheral (General disorders) | 1 (1) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0)
ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
tension headache (Nervous system disorders) | 1 (1) | 0 (0)
cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrooesophageeal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
lung neoplasm maligant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
plague shift (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
blood glucose icreased (Investigations) | 1 (1) | 0 (0)
glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Investigational Device (Test) (N=205) | PROMUS Element Plus Investigational Device (Control) (N=207)
angina pectoria (Cardiac disorders) | 17 (17) | 10 (12)
others (Cardiac disorders) | 7 (9) | 10 (12)
others (General disorders) | 42 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less